CLINICAL TRIAL: NCT01973491
Title: An Open-label, One-arm, Proof of Concept Trial to Evaluate the Safety of ATX-MS-1467 (MSC2358825A) and Its Effect on Immune Tolerance in Subjects With Relapsing Multiple Sclerosis
Brief Title: ATX-MS-1467 in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200166-001; 2013-002916-28 (EudraCT Number)
Record Dates: First submitted 2013-10-23; First posted 2013-10-31 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: ATX-MS-1467 (MSC2358825A); Relapsing Multiple Sclerosis; Magnetic resonance imaging (MRI); M2736
MeSH Terms: conditions — Multiple Sclerosis | interventions — ATX-MS-1467

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATX-MS-1467 (Experimental)
  Interventions: Drug: ATX-MS-1467

INTERVENTIONS:
Drug: ATX-MS-1467 — Subjects will receive ATX-MS-1467 50 microgram (mcg), 200 mcg and 800 mcg on Day 1, Day 15 and Day 29 respectively during the titration period followed by biweekly dose of ATX-MS-1467 800 mcg for 16 weeks during the treatment period.
  Other Names: M2736; IL-10 Inducer

SUMMARY:
This is a multi-center, open-label, single arm, baseline-controlled Phase 2a trial to evaluate the clinical and biological effects of ATX-MS-1467 in subjects with relapsing multiple sclerosis (MS) and to assess the maintenance of any such effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-patients aged 18 to 65 years of age inclusive at the time of informed consent
* Willing and able to provide written informed consent and to comply with the requirements of the protocol assessments/procedures
* Relapsing MS (relapsing-remitting multiple sclerosis [RRMS], secondary progressive multiple sclerosis [SPMS], as defined by the revised McDonald criteria [2010]) (11)
* Clinical evidence of recent MS activity and radiological activity on gadolinium (Gd)-enhanced magnetic resonance imaging (MRI) defined as defined in the protocol
* Expanded disability status scale (EDSS) score 0-5.5
* Human leukocyte antigen-beta chain (HLA-DRB)1*15 positive
* Neurological stability in the 30 days prior to Visit 5 (Study Day 1)
* Prior vaccination against tuberculosis (TB)
* If female, unless post-menopausal (for at least 2 years) or surgically sterilized, must be willing to use two highly effective methods of contraception throughout the entire duration of the trial and for 90 days following the last dose of ATX-MS-1467
* If male, must be willing to use two highly effective methods of contraception throughout the entire duration of the trial and for 90 days following the last dose of ATX-MS-1467

Exclusion Criteria:

* Primary progressive MS
* Inability to comply with MRI scanning, including contra-indications to MRI such as known allergy to gadolinium contrast dyes, claustrophobia, presence of a pacemaker, cochlear implants, ferromagnetic devices or clips, intracranial vascular clips, insulin pumps, nerve stimulators
* Previous treatment with beta-interferon, plasma exchange, intravenous gamma globulin within the 8 weeks prior to study Day 1 (Visit 5), steroids (administered via the oral and/or parenteral routes) or adrenocorticotropic hormone within the 30 days prior to the Visit 2 MRI scan, glatiramer acetate, cytotoxic agents
* Prior exposure to dimethyl fumurate (BG-12) or dirucotide, any disease-related T cell vaccine or peptide-tolerizing agent for the treatment of MS, including ATX-MS-1467
* Use of any investigational drug or experimental procedure for MS (including cytokine or anticytokine therapy) within the 30 days prior to screening (Visit 1)
* Inadequate liver function as defined in the protocol.
* Lymphocyte count less than (<)500 per micro liter (/mcL) or neutrophil count < 1500 mcL at screening or at any of the pre-treatment visits (Visits 2-4)
* Major medical illness as defined in the protocol
* Known history of active or chronic infectious disease or any disease which compromises immune function
* Any renal condition that would preclude the administration of gadolinium
* History of malignancy, including both solid tumor and hematological malignancies, but excluding basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved, in situ cervical cancer or prostatic cancer with normal prostatic specific antigen
* Clinical evidence of severe uncontrolled depression, active suicidal ideation or suicide attempt
* Any other significant medical or psychiatric conditions that, in the opinion of the Investigator, would preclude participation in the trial or impair the ability to give informed consent
* Major surgery in the 4 weeks prior to screening (Visit 1)
* Known hypersensitivity to the trial medication or diluents
* Participation in another clinical trial within the 30 days prior to screening (Visit 1)
* Pregnancy, lactation or a positive pregnancy test during screening (urine dipstick) or at Visit 4 (serum beta-human chorionic gonadotrophin [beta-hCG]), or intention to become pregnant or to breast-feed during the course of the trial
* Legal incapacity or limited legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 subjects were enrolled in the study and entered the 8-week Baseline Control Period. Following completion of the Baseline Control Period, eligible subjects entered the 4-week Titration Period followed by a 16-week Treatment Period.
Groups:
- ATX-MS-1467: Subjects received ATX-MS-1467 50 microgram (mcg), 200 mcg and 800 mcg on Day 1, Day 15 and Day 29 respectively during the titration period followed by biweekly dose of ATX-MS-1467 800 mcg for 16 weeks during the treatment period.
Period: Baseline Control Period (8 Weeks)
Arm/Group | ATX-MS-1467
Started | 37
Completed | 19
Not Completed | 18
Not completed — Did not meet Eligibility Criteria | 17
Not completed — Withdrawal by Subject | 1
Period: Titration Period(4 Weeks)
Arm/Group | ATX-MS-1467
Started | 19
Completed | 19
Not Completed | 0
Period: Treatment Period (16 Weeks)
Arm/Group | ATX-MS-1467
Started | 19
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The Safety (SAF) Analysis Set included all subjects who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- ATX-MS-1467: Subjects received ATX-MS-1467 50 mcg, 200 mcg and 800 mcg on Day 1, Day 15 and Day 29 respectively during the titration period followed by biweekly dose of ATX-MS-1467 800 mcg for 16 weeks during the treatment period.
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Number of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs) Over On-treatment Scans
Description: T1 CELs were measured using Magnetic Resonance Imaging (MRI) scans. Baseline value was calculated as the average number of T1 CELs during the 3 visits in the Baseline Control Period (Weeks -8, -4 and 0) and On-treatment value was calculated as the average number of T1 CELs during the 3 visits in the treatment period (Weeks 12, 16 and 20). The change from baseline in average number of T1 CELs was reported.
Time Frame: Baseline (Weeks -8, -4 and 0), Treatment Period (Weeks 12, 16 and 20)
Population: The modified intention-to-treat (mITT) analysis set included all enrolled subjects who received at least 1 dose of IMP and had 2 or more MRI scans during the Baseline Control Period and planned on-treatment visits (Weeks 12, 16, and 20) or end of treatment visit provided it occurred within 28 days of the last dose of IMP.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
lesions
  Baseline | 7.4 (7.62)
  Change Over Treatment Period | -2.4 (4.37)

2. Secondary Outcome: Total Number of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs)
Description: The number of T1 CELs were measured using MRI scans.
Time Frame: Weeks 12, 16, 20, 24, 28 and 36
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
lesions
  Week 12 | 3.1 (3.92)
  Week 16 | 4.6 (6.26)
  Week 20 | 5.6 (9.55)
  Week 24 | 4.9 (11.07)
  Week 28 | 2.6 (3.28)
  Week 36 | 2.2 (2.39)

3. Secondary Outcome: Change From Baseline in Total Number of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs) at Weeks 12, 16, 20, 24, 28 and 36
Description: T1 CELs were measured using MRI scans. Baseline was calculated as the average number of T1 CELs during the 3 visits in the Baseline Control Period (Weeks -8, -4 and 0).
Time Frame: Baseline (Weeks -8, -4 and 0), Weeks 12, 16, 20, 24, 28 and 36
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
lesions
  Change at Week 12 | -3.0 (4.90)
  Change at Week 16 | -2.8 (5.20)
  Change at Week 20 | -1.6 (5.11)
  Change at Week 24 | -2.2 (7.10)
  Change at Week 28 | -4.2 (7.06)
  Change at Week 36 | -4.6 (6.73)

4. Secondary Outcome: Change From Baseline in Total Volume of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs) at Weeks 12, 16, 20, 24, 28 and 36
Description: as for outcome 3
Time Frame: Baseline (Weeks -8, -4, 0), Week 12, 16, 20, 24, 28 and 36
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
milliliter
  Baseline | 0.838 (1.0151)
  Change at Week 12 | -0.321 (0.5618)
  Change at Week 16 | -0.316 (0.7184)
  Change at Week 20 | -0.225 (0.7845)
  Change at Week 24 | -0.333 (0.8622)
  Change at Week 28 | -0.454 (0.9403)
  Change at Week 36 | -0.579 (0.8807)

5. Secondary Outcome: Total Number of New or Newly Enlarging Time Constant 2 (T2) Lesions
Description: T2 lesions were measured using MRI scans.
Time Frame: Weeks 12, 16, 20, 24, 28 and 36
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
lesions
  Week 12 | 14.7 (20.69)
  Week 16 | 4.5 (6.16)
  Week 20 | 5.4 (10.07)
  Week 24 | 4.9 (8.27)
  Week 28 | 2.6 (3.28)
  Week 36 | 4.2 (3.68)

6. Secondary Outcome: Change From Week 0 in Total Number of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs) at Weeks 12, 16, 20, 24, 28 and 36
Description: T1 CELs were measured using MRI scans.
Time Frame: Week 0, 12, 16, 20, 24, 28 and 36
Population: The mITT analysis set. Here, "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure and "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 18
lesions
  Week 0 | 7.2 (6.71)
  Change at Week 12 | -3.4 (6.67)
  Change at Week 16 | -2.3 (7.03)
  Change at Week 20 | -0.9 (8.57)
  Change at Week 24 | -1.5 (10.87)
  Change at Week 28 | -3.1 (5.04)
  Change at Week 36 | -3.5 (4.40)

7. Secondary Outcome: Change From Week 0 in Total Volume of Time Constant 1 (T1) Contrast-enhanced Lesions (CELs) at Weeks 12, 16, 20, 24, 28 and 36
Description: T1 CELs were measured using MRI scans.
Time Frame: Weeks 0, 12, 16, 20, 24, 28 and 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 18
milliliter
  Week 0 | 0.815 (0.8121)
  Change at Week 12 | -0.420 (0.7520)
  Change at Week 16 | -0.264 (0.7737)
  Change at Week 20 | -0.157 (0.9839)
  Change at Week 24 | -0.271 (1.4318)
  Change at Week 28 | -0.341 (0.4541)
  Change at Week 36 | -0.473 (0.5914)

8. Secondary Outcome: Mean Annualized Relapse Rate
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. These new or worsening symptoms should be noted by the subject and must be accompanied by at least one of the following: An increase of greater than or equal to (>=) 1 grade in >=2 functional scales of the Expanded Disability Status Scale (EDSS) or an increase of >=2 grades in 1 functional scale of the EDSS or an increase of >= 0.5 or an increase of >=1.0 in EDSS if the previous EDSS was 0. Annualized Relapse Rate was calculated as = 365.25 x (Number of relapses during Treatment Period) per (Number of days on treatment during Treatment Period).
Time Frame: Week 20
Population: Analysis population included subset of mITT analysis set who had relapse.
Measure: Mean (Standard Deviation); unit: relapse per year
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 3
relapse per year | 2.60 (0.011)

9. Secondary Outcome: Time to First Relapse
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. These new or worsening symptoms should be noted by the subject and must be accompanied by at least one of the following: An increase of greater than or equal to (>=) 1 grade in >=2 functional scales of the Expanded Disability Status Scale (EDSS) or an increase of >=2 grades in 1 functional scale of the EDSS or an increase of >= 0.5 or an increase of >=1.0 in EDSS if the previous EDSS was 0. Time to first relapse was defined as the time in days from the date of first dose of study treatment to the date of first multiple sclerosis relapse.
Time Frame: Baseline up to Week 36
Population: The mITT analysis set included all enrolled subjects who received at least 1 dose of IMP and had 2 or more MRI scans during the Baseline Control Period and planned on-treatment visits (Weeks 12, 16, and 20) or end of treatment visit provided it occurred within 28 days of the last dose of IMP.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
days | NA [NA to NA] — Outcome was to be assessed as time to event analysis by Kaplan-Meier estimates. However, median and 95% CI were not estimable since very few subjects had relapse during the study.

10. Secondary Outcome: Change From Baseline in Total Expanded Disability Status Scale (EDSS) Score at Week 20
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in subjects with Multiple Sclerosis. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as any other neurological findings due to Multiple Sclerosis. Total EDSS score ranges from 0 (normal neurological examination) to 10 (death due to MS). Baseline was defined as the last measurement taken prior to the first dose of study drug (Week 0).
Time Frame: Baseline (Week 0) and Week 20
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
units on a scale
  Baseline (Week 0) | 2.32 (0.803)
  Change at Week 20 | -0.11 (0.916)

11. Secondary Outcome: Change From Baseline in Total Multiple Sclerosis Functional Composite (MSFC) Score at Week 20
Description: The MSFC is a multidimensional clinical outcome measure which consists of three sub-tests; Timed 25-Foot Walk, 9-Hole Peg Test and Paced Auditory Serial Addition Test-3(PASAT-3). The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The 9-Hole Peg Test is a quantitative measure of upper extremity (arm and hand) function. The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Standardized results (Z-scores) of these sub-tests and the overall MSFC Z-score as an average of these three Z-scores was calculated. Higher Z-scores reflect better neurological function and a positive change from baseline indicates improvement. An increase in score indicates an improvement (range -3 to +3). Baseline was defined as the last measurement taken prior to the first dose of study drug (Week 0).
Time Frame: Baseline (Week 0) and Week 20
Population: The mITT analysis set. Here, "Number Analyzed" signifies those subjects who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
Z-score
  Baseline (Week 0) | 0.001 (0.7215)
  Change at Week 20 | 0.187 (0.4321)

12. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the date of first dose and within 28 days after the date of last dose in the current study. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 25
Population: The SAF Analysis Set included all subjects who received at least 1 dose of IMP.
Measure: Number; unit: subjects
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
subjects
  TEAEs | 15
  Serious TEAEs | 0
  TEAEs Leading to Death | 0
  TEAEs Leading to Discontinuation | 1

13. Secondary Outcome: Number of Subjects Experiencing Injection Site Reactions (ISRs)
Description: Treatment-emergent ISRs were defined as any ISR with a start date on or after the date of first dose and within 7 days after the date of last dose in the current study. Injection site reactions were identified as erythema, induration, pruritus, nodules and/or cysts, ecchymosis, pain and local edema.
Time Frame: Baseline up to Week 22
Population: The SAF Analysis Set included all subjects who received at least 1 dose of IMP.
Measure: Number; unit: subjects
Arm/Group | ATX-MS-1467
Number analyzed (Participants) | 19
subjects | 7

ADVERSE EVENTS:
Time Frame: Baseline up to Week 25
Arm/Group | ATX-MS-1467
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 15/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATX-MS-1467 (N=19)
Nasopharyngitis (Infections and infestations) | 3
Cervicitis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Vaginitis gardnerella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Neutrophilia (Blood and lymphatic system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Injection site erythema (General disorders) | 5
Injection site induration (General disorders) | 2
Injection site pain (General disorders) | 2
Injection site pruritus (General disorders) | 2
Injection site haemorrhage (General disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Monocyte count decreased (Investigations) | 1
Monocyte percentage decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Reticulocyte count decreased (Investigations) | 1
Weight decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No